CLINICAL TRIAL: NCT04879225
Title: The Impact of Menthol and Mint E-liquid Bans on Menthol Cigarette Smokers
Brief Title: Menthol and Mint Experimental Tobacco Marketplace (ETM) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB00065077
Record Dates: First submitted 2021-04-13; First posted 2021-05-10 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2022-04

CONDITIONS: Cigarette Smoking; Vaping
Keywords: smoking; menthol; mint; vaping; menthol ban
MeSH Terms: conditions — Cigarette Smoking; Vaping; Smoking | interventions — Menthol; SPEN protein, human

STUDY DESIGN:
Intervention Model Description: Participants will experience four marketplace conditions that differ in the availability of flavored e-liquids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1: Fruit, dessert, mint, menthol, tobacco (Experimental): All participants receive all interventional e-liquid flavors on separate days.
  Interventions: Behavioral: All e-liquid flavors
- Intervention 2: Mint, menthol, and tobacco (Experimental): All participants receive all interventional e-liquid flavors on separate days.
  Interventions: Behavioral: Mint, Menthol and Tobacco e-liquids
- Intervention 3: Menthol and Tobacco (Experimental): All participants receive all interventional e-liquid flavors on separate days.
  Interventions: Behavioral: Menthol and Tobacco e-liquids
- Intervention 4: Only tobacco (Experimental): All participants receive all interventional e-liquid flavors on separate days.
  Interventions: Behavioral: Tobacco e-liquids

INTERVENTIONS:
Behavioral: Tobacco e-liquids — Marketplace includes tobacco flavored e-liquids
  Arms: Intervention 4: Only tobacco
Behavioral: Menthol and Tobacco e-liquids — Marketplace includes menthol and tobacco flavored e-liquids
  Arms: Intervention 3: Menthol and Tobacco
Behavioral: Mint, Menthol and Tobacco e-liquids — Marketplace includes mint, menthol and tobacco flavored e-liquids
  Arms: Intervention 2: Mint, menthol, and tobacco
Behavioral: All e-liquid flavors — Marketplace includes fruit, dessert, mint, menthol and tobacco flavored e-liquids
  Arms: Intervention 1: Fruit, dessert, mint, menthol, tobacco

SUMMARY:
Menthol cigarettes comprise almost one-third of the United States (US) market share and are disproportionately smoked by racial minorities. Tobacco control policies targeting menthol flavoring in tobacco could have significant public health outcomes, especially among black smokers. One key challenge of tobacco regulation is weighing the risks and benefits of potential policies across different populations (i.e., users and non-users). Tension arises between policies intended to prevent adolescent and young adult (AYA) tobacco initiation and those intended to reduce harm among current tobacco users. The availability of menthol e-liquids may be important for encouraging menthol cigarette smokers to switch to e- cigarettes, but mint e-liquids, which are appealing to AYA, may be unnecessary to facilitate switching. Including mint e-liquids in flavor bans but allowing menthol e-liquids to remain on the market as potential substitution products for menthol smokers may be an optimal policy approach. The study team is proposing a lab study and field assessment to determine how including menthol and mint e-liquids in e-liquid flavor bans or sales restrictions affects tobacco product purchasing and use among menthol cigarette smokers. At lab sessions, participants will complete the Experimental Tobacco Marketplace (ETM) task, a behavioral economics task in which they receive account balances to an online store and can buy menthol cigarettes at escalating costs or buy e-liquids, non-menthol cigarettes, or nicotine replacement gum at fixed costs. They will complete the task under four marketplace conditions: (1) only tobacco e-liquids available, (2) menthol and tobacco e-liquids available, (3) menthol, mint, and tobacco e-liquids available, and (4) tobacco, menthol, mint, fruit, dessert. During a field assessment, product choice is validated by assessing use of products purchased during the ETM task. This proposal will inform policy-makers about the impact banning menthol and mint e-liquids will have on facilitating menthol cigarette smokers switching to e-cigarettes.

DETAILED DESCRIPTION:
The study team proposes to conduct a within-subjects, multi-session virtual lab study and validation field assessment to determine how the availability of menthol and mint e-liquids affects product purchasing among menthol cigarette smokers. Adult daily menthol cigarette smokers will be recruited for this study. After initial eligibility is assessed, participants will complete six virtual sessions and one field assessment to evaluate their tobacco use.

Participants will be recruited from Winston-Salem, North Carolina (NC) and the surrounding area using advertisements on public transit, community flyers, and social media. Curbside visits to drop off biosamples and pickup study products will be conducted outside the Wake Forest Tobacco Control Center of Excellence located in Biotech Place in the Innovation Quarter.

The study team anticipates recruiting up to 100 participants to achieve 80 completers. Equal numbers of black and white participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. 21+ years of age
2. Self-report smoking at least 5 cigarettes per day for the past year
3. Self-report smoking menthol cigarette brands > 80% of the time
4. Breathe carbon monoxide (CO) level > 8 ppm Willingness to use other tobacco products during the study
5. Speak, comprehend, and read English sufficiently to complete study procedures
6. Have home access to a computer or tablet with a web camera and internet access

Exclusion Criteria:

1. Currently seeking treatment to quit smoking
2. Self-reported serious medical or psychiatric condition(s) including cardiovascular and chronic respiratory diseases
3. Body temperature > 100.4 F
4. Cold, flu or Novel Coronavirus (COVID-19) symptoms including fever, cough, and runny nose in the past 30 days
5. Currently pregnant, breastfeeding or intending to become pregnant for the duration of the study or unwilling to agree to use adequate protection to avoid pregnancy
6. CO reading > 80 ppm
7. Enrollment stratum (Non-Hispanic, white or Black/African American)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Denlinger, PhD, MPH, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 participants screen failed prior to enrolling.
Groups:
- E-liquid Availability: Flavor availability is manipulated
  Tobacco e-liquids: Marketplace includes tobacco flavored e-liquids
  Menthol and Tobacco e-liquids: Marketplace includes menthol and tobacco flavored e-liquids
  Mint, Menthol and Tobacco e-liquids: Marketplace includes mint, menthol and tobacco flavored e-liquids
  All e-liquid flavors: Marketplace includes fruit, dessert, mint, menthol and tobacco flavored e-liquids
Period: Fruit, Dessert, Mint, Menthol, Tobacco
Arm/Group | E-liquid Availability
Started | 52
Completed | 52
Not Completed | 0
Period: Mint, Menthol, Tobacco
Arm/Group | E-liquid Availability
Started | 52
Completed | 51
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Menthol and Tobacco
Arm/Group | E-liquid Availability
Started | 52
Completed | 51
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Only Tobacco
Arm/Group | E-liquid Availability
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Two participants were excluded from data analysis due to being unable to verify what shopping conditions the participants received.
Arm/Group | E-liquid Availability
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 44.9 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 33
  White | 17
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Combusted Tobacco Purchased
Description: Total amount of non-menthol cigarettes purchased when menthol cigarettes are not available.
Time Frame: Day 3
Population: 2 participants were excluded from data analysis due to receiving incorrect shopping links.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- E-liquid Availability: All e-liquid flavors: Marketplace includes fruit, dessert, mint, menthol and tobacco flavored e-liquids
Arm/Group | E-liquid Availability
Number analyzed (Participants) | 50
mg | 990.6 (1756.9)

2. Primary Outcome: Total Amount of Combusted Tobacco Purchased
Description: Total amount of non-menthol cigarettes purchased when menthol cigarettes are not available.
Time Frame: Day 4
Population: 2 participants were excluded from data analysis due to receiving incorrect shopping links. 1 participant was lost to follow up.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- E-liquid Availability: Mint, Menthol and Tobacco e-liquids: Marketplace includes mint, menthol and tobacco flavored e-liquids
Arm/Group | E-liquid Availability
Number analyzed (Participants) | 49
mg | 1185.9 (1510.4)

3. Primary Outcome: Total Amount of Combusted Tobacco Purchased
Description: Total amount of non-menthol cigarettes purchased when menthol cigarettes are not available.
Time Frame: Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Groups:
- E-liquid Availability: Menthol and Tobacco e-liquids: Marketplace includes menthol and tobacco flavored e-liquids
Arm/Group | E-liquid Availability
Number analyzed (Participants) | 49
mg | 1154.1 (1839.6)

4. Primary Outcome: Total Amount of Combusted Tobacco Purchased
Description: Total amount of non-menthol cigarettes purchased when menthol cigarettes are not available.
Time Frame: Day 6
Population: 2 participants were excluded from data analysis due to receiving incorrect shopping links.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- E-liquid Availability: Tobacco e-liquids: Marketplace includes tobacco flavored e-liquids
Arm/Group | E-liquid Availability
Number analyzed (Participants) | 50
mg | 1318.2 (1678.6)

5. Secondary Outcome: Total Amount of E-liquid Purchased
Description: Total amount of e-liquid purchased when menthol cigarettes are not available.
Time Frame: Day 3, Day 4, Day 5, Day 6
Population: All active participants went through all four interventions on four different days.
Measure: Mean (Standard Deviation); unit: Mg
Arm/Group | Intervention 1: Fruit, Dessert, Mint, Menthol, Tobacco | Intervention 2: Mint, Menthol, and Tobacco | Intervention 3: Menthol and Tobacco | Intervention 4: Only Tobacco
Number analyzed (Participants) | 50 | 49 | 49 | 50
Mg
  Day 3: number analyzed (Participants) | 50 | 0 | 0 | 0
  Day 3 | 9.8 (26.2) |  |  |
  Day 4: number analyzed (Participants) | 0 | 49 | 0 | 0
  Day 4 |  | 13.1 (36.4) |  |
  Day 5: number analyzed (Participants) | 0 | 0 | 49 | 0
  Day 5 |  |  | 22.4 (47.8) |
  Day 6: number analyzed (Participants) | 0 | 0 | 0 | 50
  Day 6 |  |  |  | 30.2 (56.5)

6. Other Pre Specified Outcome: Total Amount of Non-menthol Cigarettes
Description: Total amount purchased when menthol cigarettes are not available according to race
Time Frame: Day 3, Day 4, Day 5, Day 6
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Total Amount of Tobacco E-liquid Purchased
Description: Total amount of tobacco e-liquid purchased when menthol cigarettes are not available according to race.
Time Frame: Day 3, Day 4, Day 5, Day 6
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Total Amount of Menthol E-liquid Purchased
Description: Total amount of menthol e-liquid purchased when menthol cigarettes are not available according to race.
Time Frame: Day 3, Day 4, Day 5, Day 6
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Total Amount of Mint E-liquid Purchased
Description: Total amount of mint e-liquid purchased when menthol cigarettes are not available according to race.
Time Frame: Day 3, Day 4, Day 5, Day 6
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Total Amount of Dessert/Fruit E-liquid Purchased.
Description: Total amount of dessert/fruit e-liquid purchased when menthol cigarettes are not available according to race.
Time Frame: Day 3, Day 4, Day 5, Day 6
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Themes Emerging From the Qualitative Interviews
Description: Qualitative interviews will be conducted and then analyzed in an effort to learn common themes or trends among the participants specific to various tobacco and nicotine products.
Time Frame: Day 14
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mean Perceived Health Risk Scale Score
Description: This is a measure of the perceived addictive potential and other health risks associated with cigarettes, e-cigarettes and nicotine gum. Scale 1-10 (1=very low risk of disease and 10=very high risk of disease). Each item/question has a score of 1-10. There are 14 different items in this questionnaire and each item will be evaluated independently.
Time Frame: Baseline, Day 14
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mean Product Evaluation Scale Score
Description: This scale measures the participant's experience while using cigarettes, nicotine gum, or vaping devices. Each of the three products will include 13 items with a total score range of 13-91 for each of the three products. A higher score denotes more enjoyment from the product.
Time Frame: Baseline, Day 14
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mean Minnesota Nicotine Withdrawal Scale Score
Description: This is a 15-item self-reported scale to evaluate the effects of smoking cessation and withdrawal symptoms. This scale is important because it allows the researchers to understand the experience of the participant throughout the study while using various tobacco products. The study team will use 7/15 items from this scale each ranging in score from 1-5. Total score range for the questionnaire would be 7-35 with higher score denoting more severe symptoms.
Time Frame: Baseline, Day 3, Day 4, Day 5, Day 6, Day 14
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Mean Questionnaire on Smoking Urges Score
Description: This scale measures the person's urge to smoke throughout the study while potentially using various tobacco and nicotine products. This questionnaire consists of 10 items each ranging from 1-7. Total score range for the entire questionnaire is 10-70. A higher score denotes greater urge.
Time Frame: Baseline, Day 3, Day 4, Day 5, Day 6, Day 14
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Mean Tobacco Product Interest Scores
Description: A visual analog scale assessing interest in use of various tobacco and nicotine products. Each item has a score from 0-100. This scale ranges from no interest (0) to very interested (100). The total questionnaire has 9 items that will be evaluated independently. The study team is looking at the following:
  1. Preferred cigarette brand
  2. Any other cigarette brand
  3. A cigarette brand with 95% less nicotine
  4. I Quit Ordinary Smoking (IQOS) Heat-Not-Burn Device
  5. Juice Universal Serial Bus Lighting (JUUL) Vaping Device
  6. Zyn Nicotine Pouches
  7. NicoDerm Nicotine Patch
  8. Nicorette Nicotine Lozenge
  9. Nicorette Nicotine Gum
Time Frame: Baseline, Day 14
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Tobacco Policy Questionnaire Score
Description: A visual analog scale assessing interest in use of various tobacco and nicotine products. This questionnaire will assess support for various tobacco control policies, including banning menthol flavoring in cigarettes and e-cigarettes. Each of the 14 items has a score of 1-3. 1 means the subject is supportive of the policy, 2 means subject is opposed. 3 indicates that the subject does not know. Each of the 14 items will be evaluated independently from one another.
Time Frame: Baseline, Day 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through Day 14
Arm/Group | E-liquid Availability
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

LIMITATIONS AND CAVEATS:
Several recruitment methods were utilized to identify participants including flyers, Craigslist and contracting with a clinical research recruitment agency. All methods yielded participants but ultimately were not enough to meet our enrollment goal of 80 participants. We experienced a significant uptick in the number of enrolled participants in the final months of the study. We attribute this to the temporal change that has resulted from a return to normal activities after the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT04879225/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04879225/ICF_002.pdf